CLINICAL TRIAL: NCT05202743
Title: Cultivating Self-Compassion Course for Persons Living With Amyotrophic Lateral Sclerosis
Brief Title: Online Self-Compassion Course for pALS (Compassion pALS)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202110073
Record Dates: First submitted 2021-12-29; First posted 2022-01-21 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational for ALS patients — Open to ALS patients interested in mindfulness training.

SUMMARY:
This study is designed to be a pragmatic, single-arm trial to evaluate the efficacy, implementation, and feasibility of an online ALS-specific self-compassion training program to enhance self-compassion and improve quality of life.

DETAILED DESCRIPTION:
Optimizing quality of life for people with ALS is a primary goal of ALS multidisciplinary care, Therefore, it is especially important to conduct research into interventions to address the psychological needs and well-being of people with ALS.

Recent studies have shown that mindfulness-based interventions promote improved quality of life for people with ALS. It is essential that such strategies as mindfulness-based interventions consider the specific needs of the ALS population and potential barriers to participation.

Very few studies have evaluated mindfulness-based interventions in the ALS population and no studies to date have evaluated self-compassion people with ALS. Self-compassion has been linked to increased emotional resilience, psychological well-being, and quality of life in multiple populations.

The intervention will include a 2-part workshop entitled 'Introduction to Mindful Self-Compassion for Persons Living with Amyotrophic Lateral Sclerosis.' Experience and feedback gained from the workshop will be incorporated into the format for an 8-week course in Cultivating Self-Compassion for persons living with ALS (Compassion pALS). Compassion pALS will be adapted from the Mindful Self-Compassion (MSC) Program to accommodate ALS clinical features and limit potential barriers to participation.

The primary outcome will be quality of life assessed with the Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSA-5). Participants will be assessed at the 2-part workshop (T0, baseline), start of the 8 week Compassion pALS course (T1 = pre-intervention); after completing the intervention (T2, post-intervention). Secondary outcomes will include Secondary outcome measures the Self-Compassion Scale Short Form (SCS-SF), Patient Health Questionnaire-9 (PHQ-9), General Anxiety Disorder-7 (GAD-7), Amyotrophic Lateral Sclerosis Functional Rating Scale-R (ALSFRS-R), Feasibility of Intervention Measure (FIM), Acceptability of Intervention Measure (AIM), and Intervention Appropriateness Measure (IAM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS within the last 18 months.
* 18 years or older
* Access to and the physical ability to use a computer with internet access with and/or without adaptive devices.
* Ability to communicate and understand tasks.
* A caregiver available to provide assistance.
* Ability to provide informed consent

Exclusion Criteria:

* More than one neuropsychological impairment such as (frontotemporal dementia) which may interfere with the study procedures.
* Severe medical condition that would reduce life expectancy to less than 6-12 months.
* No access to a computer with internet access
* Unsuitable for the study as determined by the Investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ALS participants will be recruited from a Neuromuscular clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life self-assessment with - Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSA-5) | Baseline (T1); post 8-week intervention (T2)
  Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSAQ-5; Jenkinson et al., 2001.

SECONDARY OUTCOMES:
Self-compassion | Baseline (T1); post 8-week intervention (T2)
  Self-Compassion Scale Short Form (SCS-SF; Raes et al., 2011)
Participant functional rating self-assessment | Baseline (T1); post 8-week intervention (T2)
  Self-Administered ALS Functional Rating Scale-Revised (SA-ALSFRS; Montes et al., 2006)
Anxiety | Baseline (T1); post 8-week intervention (T2)
  General Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006)
Depression | Baseline (T1); post 8-week intervention (T2)
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2002)
Feasibility of implementation | Baseline (T1); post 8-week intervention (T2)
  Feasibility of Intervention Measure (FIM; Weiner et al., 2017)
Acceptability | Baseline (T1); post 8-week intervention (T2)
  Acceptability of Intervention Measure (AIM; Weiner et al., 2017)
Appropriateness | Baseline (T1); post 8-week intervention (T2)
  Intervention Appropriateness Measure (IAM; Weiner et al., 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Smith, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States